CLINICAL TRIAL: NCT03308864
Title: Strong Connections-Interpersonal Psychotherapy for Adolescents
Brief Title: Strong Connections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Elizabeth Handley, Research Associate, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB44140
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal Psychotherapy for Adolescents (IPT-A) (Experimental): All adolescents who present at Child and Adolescent Outpatient Service (CAOS) for a diagnostic intake evaluation and who report any symptoms of depression.
  Interventions: Behavioral: Interpersonal Psychotherapy for Adolescents
- Treatment as Usual (Active Comparator): All adolescents who present at Child and Adolescent Outpatient Service (CAOS) for a diagnostic intake evaluation and who report any symptoms of depression.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Adolescents — Experimental: Interpersonal Psychotherapy for Adolescents (IPT-A) IPT-A is a manualized intervention for depression that targets adolescents' interpersonal context and social supports as mechanisms of change. It will be provided in accordance with the treatment manual by Child and Adolescent Outpatient Service clinicians over the course of 12-16 50-minute sessions.
  Arms: Interpersonal Psychotherapy for Adolescents (IPT-A)
Behavioral: Treatment as usual — Treatment as usual will consist of the standard care for adolescent depressive symptoms at CAOS. TAU is not manualized; it is consistent with care typically provided in community settings. Therapists establish a working alliance, are empathetic, reflect expressed affect, and discuss options for coping with concerns as initiated by the adolescent.
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to compare two talking forms of therapy designed to help reduce depressive symptoms in teenagers: Interpersonal Psychotherapy for Adolescents and Treatment as Usual.

DETAILED DESCRIPTION:
Interpersonal Psychotherapy for Adolescents (IPT-A) is a manualized short-term therapeutic intervention that has been shown to be efficacious in a number of randomized control trials for adolescent depression. The primary aim of the present study is to evaluate the feasibility of incorporating Interpersonal Psychotherapy for Adolescents (IPT-A) into routine psychotherapeutic treatment at Strong Behavioral Health: Child and Adolescent Outpatient. The second aim of the present investigation is to examine changes in adolescent symptomatology, interpersonal functioning, perceived stress, and social support throughout the course of treatment. The third aim of the present study is to compare the effectiveness of IPT-A versus treatment as usual (TAU) at reducing depressive symptoms among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* age 12-18
* scoring in the clinically elevated range for depression using the Beck Depression Inventory for Youth

Exclusion Criteria:

* currently psychotic
* do not speak English
* currently participating in another form of mental health treatment
* considered to need inpatient hospitalization
* IQ less than 70

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Mean Beck Depression Inventory score | Baseline to 8 months
  Adolescents' depressive symptomatology will be measured using adolescent-report of the Beck Depression Inventory-Youth. It is a 20-item scale ranging from 0 to 100 with higher scores indicating worse health outcomes.
Change in Mean Beck Depression Inventory score | Baseline to 5 months
  Adolescents' depressive symptomatology will be measured using adolescent-report of the Beck Depression Inventory-Youth. It is a 20-item scale ranging from 0 to 100 with higher scores indicating worse health outcomes.

SECONDARY OUTCOMES:
Change in the mean score in suicide ideation. | Baseline to 5 months
  The Beck Suicide Scale will be used to measure suicide ideation. It is a 21-item scale ranging from 0-2 with higher scores higher levels of suicide ideation.
Change in the mean score in suicide ideation. | Baseline to 8 months
  The Beck Suicide Scale will be used to measure suicide ideation. It is a 21-item scale ranging from 0-2 with higher scores higher levels of suicide ideation.
Change in mean perceived stress | Baseline to 5 months
  The Perceived Stress Scale will be used to measure perceived stress. It is a 14-item scale ranging from 0-4 with higher scores higher levels of stress.
Change in mean perceived stress | Baseline to 8 months
  The Perceived Stress Scale will be used to measure perceived stress. It is a 14-item scale ranging from 0-4 with higher scores higher levels of stress.
Change in mean social adjustment | Baseline to 5 months
  The Social Adjustment Scale-SR will be used to measure social adjustment. It is a 23-item scale ranging from 0-5 with higher scores higher levels of social adjustment.
Change in mean social adjustment | Baseline to 8 months
  The Social Adjustment Scale-SR will be used to measure social adjustment. It is a 23-item scale ranging from 0-5 with higher scores higher levels of social adjustment.
Mean change in social support | Baseline to 5 months
  The Social Support Behaviors Scale will be used to measure social support. There are two domains, one for family and one for friends. It is a 45-item scale ranging from 0-5 with higher scores indicating higher levels of social support.
Mean change in social support | Baseline to 8 months
  The Social Support Behaviors Scale will be used to measure social support. There are two domains, one for family and one for friends. It is a 45-item scale ranging from 0-5 with higher scores indicating higher levels of social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Behavior Health and Wellness, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No